CLINICAL TRIAL: NCT05251233
Title: Evaluation of the Role of Proton Pump Inhibitors on the Postoperative Course Following Pancreaticoduodenectomy
Brief Title: Role of Proton Pump Inhibitors on the Postoperative Course Following Pancreaticoduodenectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator and study team chose to end study early.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202201171
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Ampullary Cancer; Pancreas Neuroendocrine Tumor; Pancreatitis; Distal Extrahepatic Cholangiocarcinoma; Duodenal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Duodenal Neoplasms | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): -Visually equivalent placebo once daily from postoperative day 1 and continued for 10 doses or until the day of discharge (whichever is earlier).
  Interventions: Drug: Placebo
- Proton pump inhibitor (Active Comparator): -Pantoprazole once daily from postoperative day 1 and continued for 10 doses or until the day of discharge (whichever is earlier).
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Placebo — Placebo capsules contain pharmaceutical-grade lactose monohydrate NF, a naturally occurring disaccharide of galactose bound to glucose.
  Arms: Placebo
Drug: Pantoprazole — The study will use commercial supply.
  Arms: Proton pump inhibitor

SUMMARY:
The purpose of this study is to prospectively determine the effects of administering proton pump inhibitors (PPIs) following pancreaticoduodenectomy on postoperative outcomes. The findings of this study will help in avoiding the widespread use of PPIs during the immediate postoperative period following pancreatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who will undergo pancreaticoduodenectomy with gastric/biliary reconstruction performed as definitive management for a benign or malignant disease at Washington University/Barnes-Jewish Hospital.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leigh-Matijakovich, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Unassigned Arm: For patients who were enrolled but did not get randomized or receive any treatment.
Period: Overall Study
Arm/Group | Placebo | Proton Pump Inhibitor | Unassigned Arm
Started | 21 | 20 | 15
Completed | 14 | 16 | 0
Not Completed | 7 | 4 | 15
Not completed — Disease progression - did not start treatment | 0 | 0 | 5
Not completed — Determined to be ineligible - did not start treatment | 0 | 0 | 7
Not completed — Patient was NPO with NGT, could not receive oral medication - did not start treatment | 0 | 0 | 1
Not completed — Had a total gastrectomy - did not start treatment | 0 | 0 | 1
Not completed — Death - did not start treatment | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Other complicating disease | 2 | 1 | 0
Not completed — Attending physician did not order medication for patient - did not start treatment | 0 | 0 | 1
Not completed — Patient was ordered NPO and had NGT placed. | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Proton Pump Inhibitor | Unassigned Arm | Total
Number analyzed (Participants) | 21 | 20 | 15 | 56
Age, Continuous [Median (Full Range); unit: years] | 69 [24 to 87] | 67.5 [37 to 88] | 62 [48 to 80] | 67 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 6 | 24
  Male | 12 | 11 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 15 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 20 | 20 | 15 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 15 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delayed Gastric Emptying as Measured by the International Study Group of Pancreatic Surgery (ISGPS) Criteria
Description: -Will be coded as yes and no
Time Frame: Through 90 days after surgery
Population: Three participants who were randomized to the Placebo arm died prior to receiving any treatment and are not included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Proton Pump Inhibitor
Number analyzed (Participants) | 18 | 20
Participants | 3 | 6

2. Primary Outcome: Number of Participants With Delayed Gastric Emptying as Measured by Modified Accordion Grading System (MAGS)
Description: -Will be coded as yes and no
Time Frame: Through 90 days after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Proton Pump Inhibitor
Number analyzed (Participants) | 18 | 20
Participants | 3 | 6

3. Secondary Outcome: Number of Participants With Surgical Complication(s) Defined by the Modified Accordion Grading System (MAGS)
Description: Surgical complication is defined by the Modified Accordion Grading System, coded as yes and no.
Time Frame: Through 90 days after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Proton Pump Inhibitor
Number analyzed (Participants) | 18 | 20
Participants | 8 | 11

4. Secondary Outcome: Kaplan-Meier Estimated 90-days Marginal Ulcer-free Survival (MUFS) Probability
Description: -MUFS is defined as the days from the date of randomization to diagnosis of a marginal ulcer. The patients without marginal ulcer are censored at the date of last follow-up.
Time Frame: Through 90 days after surgery
Measure: Number (95% Confidence Interval); unit: proportion probability
Arm/Group | Placebo | Proton Pump Inhibitor
Number analyzed (Participants) | 13 | 16
proportion probability | 0.9230769 [0.5663595 to 0.9887941] | 0.875 [0.5859814 to 0.9671888]

ADVERSE EVENTS:
Time Frame: - Adverse events were collected from start of treatment through 30 days after last day of PPI/placebo (up to 40 days). - All-cause mortality was collected from enrollment through 90 days after surgery (up to 90 days).
Description: * Adverse events that are considered surgical complications and are unrelated to treatment with PPI/placebo are only collected for the secondary outcome measure of surgical complications and are not presented in the adverse event module.
  * Adverse events were not collected on those participants who were in the unrandomized arm. Those participants were enrolled but were never randomized to PPI or placebo.
Arm/Group | Placebo | Proton Pump Inhibitor | Unassigned Arm
All-Cause Mortality (participants affected / at risk) | 3/21 | 0/20 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05251233/Prot_SAP_000.pdf